CLINICAL TRIAL: NCT02668263
Title: Randomised Clinical Trial Investigating the Use of Drains and Quilting Sutures on Seroma Formation Following Mastectomy - A Pilot Study
Brief Title: Investigating the Use of Drains and (Internal) Quilting Sutures on Seroma Formation Following Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Tees and Hartlepool NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Gateshead Health NHS Foundation Trust (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr Pud Bhaskar, Consultant General and Breast Oncoplastic Surgeon, North Tees and Hartlepool NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NorthTeesNHS; RECRef:14/NE/0091 R&D SUR094 (Other: NorthTeesNHS)
Record Dates: First submitted 2016-01-18; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; mastectomy; seromas
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Surgery and Drain (Active Comparator): Group 1 will be allocated to receive a drain intra-operatively.
  Interventions: Procedure: Surgery and Drain(s)
- Surgery alone (Other): Group 2 will not receive a drain and no further intervention.
  Interventions: Procedure: Surgery alone
- Surgery and quilting sutures (Experimental): Group 3 will not receive a drain but will receive quilting sutures
  Interventions: Procedure: Surgery and Quilting Sutures

INTERVENTIONS:
Procedure: Surgery alone — Surgery
  Arms: Surgery alone
Procedure: Surgery and Drain(s) — Drains inserted as per standard practice
  Arms: Surgery and Drain
Procedure: Surgery and Quilting Sutures — Quilting sutures to mastectomy flaps
  Arms: Surgery and quilting sutures

SUMMARY:
Seroma formation is a common complication following breast and axillary surgery for breast cancer. The use of drains is commonplace in practice after mastectomy, although there is evidence to suggest that they do not affect the incidence of symptomatic seroma formation. Methods have been adopted in attempts to decrease seroma formation, to varying results, which include the use of deep sutures. The aim of this study is to evaluate the effect of drains and quilting sutures on the incidence of seroma formation. Patients undergoing mastectomy and axillary surgery for breast cancer will be eligible. Patients will be randomized to either receive a drain, no drain or no drain with quilting sutures. The primary outcome measure will be the incidence of symptomatic seroma. Secondary outcome measures will be postoperative length of stay and postoperative pain scores.

DETAILED DESCRIPTION:
Background: The mainstay of treatment for the majority of breast cancers is surgical excision of the primary tumour either by removing the lump (wide local excision) or the whole breast, mastectomy. Breast cancer can commonly spread to the lymph nodes in the armpit (axilla) meaning surgery to remove the cancer also involves surgery to axilla to sample lymph nodes. The most common complication following mastectomy is a fluid collection deep to the wound called a seroma. This is generally a minor complication but may cause significant discomfort / distress to the patient. If the seroma is of a significant size as to cause discomfort, it is usually drained using a needle and syringe near the wound. This is not only to improve patient discomfort, but seromas can lead to wound healing problems which may delay the onset of adjuvant treatment, such as radio- or chemotherapy. The incidence of seroma is variable, but the most commonly quoted incidence of seroma formation is between 15% and 27%.

In a bid to reduce seroma formation, surgeons use drains following mastectomy to theoretically remove any excess fluid that may accumulate following surgery. This is the current practice in our unit at North Tees. Despite the widespread use of drains following mastectomy, there is no clear evidence to suggest that the use of drains significantly reduces seroma formation. There are also no consensus guidelines for the use of postoperative drains. Most surgeons advocate the removal of drains when the volume drained is less than 50ml/day. Patients with a drain in-situ may be kept as inpatients until drain removal, others may go home with drains with frequent review at home by the breast care nursing team. As a consequence, drains may contribute to a longer postoperative stay and have also been linked to higher postoperative pain scores.

The nature and behaviour of seromas remains ambiguous; it is hard predicting which patients will be troubled by them. There is one argument however, that seroma fluid may be increased by the presence of a drain. This is because the drain may irritate the tissues underneath the wound, resulting in the tissues producing more fluid which may accumulate into a seroma. Therefore, there lies a theoretical basis for which drains should be avoided altogether.

Other measures have been adopted other than drains in a bid to reduce seroma formation. One of the main ones are the use of 'quilting sutures' deep to the wound. These have previously been used either in addition to a drain or without. Quilting sutures aim to reduce the 'free space' left in the tissues following removal of the breast by adhering the tissues together. The free space, commonly called 'dead space' is a risk factor for the accumulation of fluid. It has been shown in studies that with or without a drain, these sutures (or stitches) reduce the incidence of seroma and reduce the length of inpatient stay.

Aim/Objective: This pilot study aims to determine the effect that drains and quilting sutures have on the incidence of symptomatic seroma formation following mastectomy and axillary surgery for breast cancer. A symptomatic seroma is defined as a fluid collection beneath the mastectomy wound which develops post-operatively, causing tension on the healing wound and discomfort to the patient, thus needing drainage. This is usually approximately 100mls or greater in quantity of fluid.

Outcome measures: See below

Population

Eligibility Criteria: see below

Sample size: This is a feasibility study which will recruit patients from four NHS Foundation Trusts in the North-East of England (North Tees and Hartlepool, Northumbria, Gateshead and Newcastle Hospitals). The principle research centre will be North Tees. No power calculation has been used to determine sample size. A small sample will be used to assess the feasibility of the intervention with the aim of using this study as a pilot for a large study in the future which would have a sample based on power calculations. Seroma incidence has been quoted as around 15-27%.2 University Hospital of North Tees and Hartlepool alone treat approximately 500 patients diagnosed with breast cancer every year. Each centre will recruit 30 patients, which approximates to 10 per group. This gives a total sample size of 120 patients.

Subjects will be recruited at the breast clinic when consenting for surgery. They will be approached regarding the study as part of the consent process.

Randomisation process: Block randomisation using computer generated opaque sealed envelopes sequencing stratified by the centre. Variable block sizes are preferable but not necessary given the three arms of the study and multiple study sites. According to site, participants will be labelled in four blocks of 30 for randomisation to make sure all sites allocate 10 in each group. These will be labelled A1-30 to D1-30. The reasoning for this method is that if participants were labelled 1-120, then there would be a need for someone who always had access to the next randomisation group. As this is a pilot study, there would not be the facility to have a 24-hour randomisation call-line. Participants will be allocated into either groups 1, 2 or 3 (as detailed below in 'Study Procedure').

Informed written consent: Consent for the study will be taken at the time of consenting for surgery at the breast clinic. This will be undertaken on a specific consent form. The patients will also be given an information leaflet at this time, with the option of returning to another clinic and consenting later.

Study Procedure: Patients eligible and who consent to be subjects in the study will be randomized into one of three groups and will receive treatment at the hospital at which they present. Pre-operative practice and operative technique will be standardised between sites and will be routine practice. Group 1 will be allocated to receive a drain intra-operatively. Group 2 will not receive a drain and no further intervention. Group 3 will not receive a drain but will receive quilting sutures. A sealed envelope will be opened by the theatre nursing staff immediately before wound closure to reveal the randomisation code. Patients in group 2 and 3 and breast care nurses will be blinded regarding the use of quilting sutures. Surgery will be carried out by consultants or experienced registrars.

Subjects in group 1 will be discharged from hospital when ambulatory and pain is controlled by oral analgesia. They may go home with the drain in-situ or be discharged when the drain is removed. The drain in either case will be removed when the output is less than 50ml in 24h. Patients in group 2 and 3 will be discharged when ambulatory and similarly analgesic requirements are met with oral preparations.

Patients will be followed up in the breast clinic in two weeks post surgery.

Those randomised to not receive a drain (Groups 2 and 3) are not anticipated to have a longer postoperative inpatient stay. On the contrary, it is anticipated they may be discharged sooner than those in group 1.

End of the study: The end of the study will be marked when subjects' seromas cease to be symptomatic or needing drainage. Participants will be followed up routinely within the breast clinic as part of their on-going cancer management.

Assessment of safety: No additional toxicity data will be required to be included. Any adverse events or safety issues will be dealt with in accordance with standard hospital protocol.

Subject withdrawal: Patients will be free to withdraw from the study at any time. This may be defined as pre or post intervention. The reasons for withdrawal will be noted in the patient records.

Data recording: Each patient will be assigned a case report form. The patient will be reviewed at 24h post-operatively and data collected by the clinician. At 24h, data on the drainage volumes in the drain group, pain scores and an examination of the wound will be conducted. Pain scores at 48h by the same scoring system will also be used. Pain scores will be recorded using a validated visual analogue score (VAS). The patient will be reviewed each day in hospital until discharge. Upon discharge, the breast care nurses will collect data on seroma incidence, aspiration volumes and wound care. Data will then be entered into a secure hospital-based Microsoft Excel spreadsheet. Transfer of data will be via NHS.net to NHS.net email to ensure security.

Statistical considerations: This is a pilot study so only requires small patient numbers therefore descriptive statistics only will be used.

Source data/documents/confidentiality: The Data Protection Act, NHS Research Governance Framework and relevant NHS codes of practice will be followed with regards to the collection, storage, processing and disclosure of personal and study information.

Participants will be given a study number at the onset of the trial, with a link to their personal data on a separate database. The main data will only be collected in reference to the unique study number and thus data will be anonymised and kept confidential.

Data will be collected on case report forms. This will then be entered into a secure hospital-based spreadsheet. The researchers will have access to the data. No patient identifiable details will be removed from the hospital site. All paper copies will be filed in a hospital-based master research file. The patient consent form will be filed in the subjects' hospital records.

As this will be a four-centre study, data will be transferred from the other sites to North Tees however no patient identifiable information will be transferred only study reference number. Transfer will be between secure NHS.net email accounts and data will be held for 5 years.

Quality control & quality assurance: This is a low risk trial and no major issues are anticipated. A formal data monitoring committee is not needed.

Either Consultant Surgeons or highly skilled specialist registrars will carry out the surgery. Patients will be closely followed up by the surgical team or breast care nurses and have open access to the breast care service. If however high complication rates are experienced in a particular group, this method will be stopped.

Quality control will be maintained by strict adherence to the study protocol, the principles of GCP, research governance and clinical trial regulations.

Ethical considerations : The main ethical issue surrounding this trial is that two thirds of patients will not receive the current practice at the four trusts, of receiving a drain. However, this is not to suggest that by not receiving a drain, they will have a less favourable outcome. The main risk to patients is a symptomatic seroma, which may require drainage. However, patients are at risk of seromas whether they have a drain put in or not, and by actually not receiving a drain, may have a lower incidence of seroma, less pain and time in hospital.

There will be strict compliance with the principles of the Declaration of Helsinki and MRC/ICH good clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Females presenting with newly diagnosed carcinoma of the breast with or without axillary node clearance or sampling.
* They must be at least 18 years of age and have capacity to give informed consent.

Exclusion Criteria:

* Male
* Those who do not have capacity
* Previous breast cancer in the same breast and previous axillary surgery
* Previous chest wall radiotherapy
* Patients with metastatic cancer including lymphoma, pre-existing lymphoedema
* Intercurrent infection or hypoalbuminaemia (<36 g/L)
* Patients part of other research trials.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Seroma formation | One week post-operatively
  Incidence of symptomatic seroma post-operatively. A seroma defined as a palpable fluid collection under the wound.

SECONDARY OUTCOMES:
Seroma aspiration | up to 1 month
  Any symptomatic seromas will be aspirated, and the volume in milliliters will be recorded.
Pain scores | up to 2 days post-operatively
  Daily Post-operative pain scores using visual analogue scale
Length of Stay | up to 1 week
  Postoperative length of stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Pud Bhaskar, MBBS, MD, Principal Investigator — North Tees & Hartepool NHS Foundation Trust
Locations (1):
- Department of Surgery, North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees, Cleveland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal A, Ayantunde AA, Cheung KL. Concepts of seroma formation and prevention in breast cancer surgery. ANZ J Surg. 2006 Dec;76(12):1088-95. doi: 10.1111/j.1445-2197.2006.03949.x. PMID 17199696
- [Background] Woodworth PA, McBoyle MF, Helmer SD, Beamer RL. Seroma formation after breast cancer surgery: incidence and predicting factors. Am Surg. 2000 May;66(5):444-50; discussion 450-1. PMID 10824744
- [Background] Hashemi E, Kaviani A, Najafi M, Ebrahimi M, Hooshmand H, Montazeri A. Seroma formation after surgery for breast cancer. World J Surg Oncol. 2004 Dec 9;2:44. doi: 10.1186/1477-7819-2-44. PMID 15588301
- [Background] Sampathraju S, Rodrigues G. Seroma formation after mastectomy: pathogenesis and prevention. Indian J Surg Oncol. 2010 Dec;1(4):328-33. doi: 10.1007/s13193-011-0067-5. Epub 2011 Apr 2. PMID 22693384
- [Background] Akinci M, Cetin B, Aslan S, Kulacoglu H. Factors affecting seroma formation after mastectomy with full axillary dissection. Acta Chir Belg. 2009 Jul-Aug;109(4):481-3. doi: 10.1080/00015458.2009.11680464. PMID 19803259
- [Background] Jain PK, Sowdi R, Anderson AD, MacFie J. Randomized clinical trial investigating the use of drains and fibrin sealant following surgery for breast cancer. Br J Surg. 2004 Jan;91(1):54-60. doi: 10.1002/bjs.4435. PMID 14716794
- [Background] Barwell J, Campbell L, Watkins RM, Teasdale C. How long should suction drains stay in after breast surgery with axillary dissection? Ann R Coll Surg Engl. 1997 Nov;79(6):435-7. PMID 9422871
- [Background] Kopelman D, Klemm O, Bahous H, Klein R, Krausz M, Hashmonai M. Postoperative suction drainage of the axilla: for how long? Prospective randomised trial. Eur J Surg. 1999 Feb;165(2):117-20; discussion 121-2. doi: 10.1080/110241599750007289. PMID 10192568
- [Background] Bailey SH, Oni G, Guevara R, Wong C, Saint-Cyr M. Latissimus dorsi donor-site morbidity: the combination of quilting and fibrin sealant reduce length of drain placement and seroma rate. Ann Plast Surg. 2012 Jun;68(6):555-8. doi: 10.1097/SAP.0b013e318216b65c. PMID 21629082
- [Background] Dancey AL, Cheema M, Thomas SS. A prospective randomized trial of the efficacy of marginal quilting sutures and fibrin sealant in reducing the incidence of seromas in the extended latissimus dorsi donor site. Plast Reconstr Surg. 2010 May;125(5):1309-1317. doi: 10.1097/PRS.0b013e3181d4fb68. PMID 20440152
- [Background] Sakkary MA. The value of mastectomy flap fixation in reducing fluid drainage and seroma formation in breast cancer patients. World J Surg Oncol. 2012 Jan 11;10:8. doi: 10.1186/1477-7819-10-8. PMID 22236813
- [Background] Schuijtvlot M, Sahu AK, Cawthorn SJ. A prospective audit of the use of a buttress suture to reduce seroma formation following axillary node dissection without drains. Breast. 2002 Feb;11(1):94-6. doi: 10.1054/brst.2001.0366. PMID 14965653